CLINICAL TRIAL: NCT05975567
Title: Deploying Novel Imaging Modalities Towards a Three-dimensional (3D) CARDIOvascular PATHology: the 3D-CARDIOPATH Study
Brief Title: Deploying Novel Imaging Modalities Towards a Three-dimensional (3D) CARDIOvascular PATHology
Acronym: 3D-CARDIOPATH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: National and Kapodistrian University of Athens (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, Andreas S Papazoglou, MD, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: 5039/69589
Record Dates: First submitted 2023-07-05; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease; Aortic Valve Calcification; STEMI; Cardiovascular Pathology
Keywords: micro-CT; light sheet fluorescence microscopy; intravascular ultrasound; optical coherence tomography; 3D cardiovascular imaging; 3D cardiovascular pathology
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease; Aortic Valve, Calcification of; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Our study aims to collect:
  1. 20 cadaveric coronary artery segments collected from 10 adults with sudden cardiac death (SCD);
  2. 30 thrombotic specimens aspirated during percutaneous coronary intervention (PCI) procedures in patients with ST-elevated myocardial infarction (STEMI);
  3. 30 calcific aortic valves surgically removed from patients with CAVD undergoing cardiac surgery for valve replacement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diseased cadaveric coronary arteries from individuals with sudden cardiac death: Cadaveric coronary artery segments (5-15 mm) will be excised at necropsy (post mortem) from 10 individuals with SCD likely to have advanced coronary atherosclerosis.
  Interventions: Other: Three-dimensional imaging of the collected cardiac specimens
- Aspirated thrombotic specimens from patients with ST-elevated myocardial infarction: Thrombotic samples will be aspirated from 30 patients with STEMI admitted to the Hippokrateion Hospital of Thessaloniki, Greece and undergoing primary PCI and routine thrombus aspiration per standardized procedures.
  Interventions: Other: Three-dimensional imaging of the collected cardiac specimens
- Calcific aortic valves surgically resected from patients with calcific aortic valve disease: Calcific aortic valves will be surgically removed from 30 patients with CAVD undergoing cardiac surgery for aortic valve replacement.
  Interventions: Other: Three-dimensional imaging of the collected cardiac specimens

INTERVENTIONS:
Other: Three-dimensional imaging of the collected cardiac specimens — The cadaveric coronary artery segments will first be scanned with intravascular imaging modalities, namely optical coherence tomography (OCT) and intravascular ultrasound (IVUS), and then with micro-computed tomography (micro-CT) and light sheet fluorescence microscopy (LSFM). The thrombotic specimens aspirated from patients with ST-elevated myocardial infarction, will also be scanned using micro-CT. The surgically removed aortic valves will undergo scanning with micro-CT and LSFM. Traditional histopathological assessment will also be performed on the scanned specimens.

SUMMARY:
The goal of the 3D-CARDIOPATH study is to investigate the potential added value of emerging 3D imaging modalities by imaging ex vivo cardiac specimens (diseased coronary arteries, calcific aortic valves, and thrombotic materials) in 3D. Specifically, 20 cadaveric coronary artery segments with advanced atherosclerosis will be received from 10 patients with SCD. These segments will first be scanned with intravascular imaging modalities, namely optical coherence tomography (OCT) and intravascular ultrasound (IVUS), and then with micro-computed tomography (micro-CT) and light sheet fluorescence microscopy (LSFM). Additionally, 30 thrombotic specimens aspirated from patients with ST-elevated myocardial infarction, will also be scanned using micro-CT. Finally, 30 surgically removed aortic valves will undergo scanning with micro-CT and LSFM. Traditional histopathological assessment will also be performed on the scanned specimens. Patient laboratory profiles, past medical histories, demographic characteristics, and therapeutic management will be recorded, where applicable.

DETAILED DESCRIPTION:
The 3D-CARDIOPATH study aims to provide 3D volumetric insights into well-characterized disease entities such as Coronary artery disease (CAD) and calcific aortic valvular disease (CAVD). Therefore, this study aims to visualize in 3D:

1. cadaveric coronary artery samples collected from adults with sudden cardiac death (SCD);
2. thrombotic specimens aspirated during percutaneous coronary intervention (PCI) procedures in patients with ST-elevated myocardial infarction (STEMI); and
3. calcific aortic valves surgically removed from patients with CAVD undergoing cardiac surgery for valve replacement.

The utilized 3D imaging means will be:

1. optical coherence tomography (OCT), intravascular ultrasound (IVUS), micro-computed tomography (micro-CT) and light sheet fluorescence microscopy (LSFM) for the assessment of the collected cadaveric coronary arteries;
2. micro-CT for the assessment of the aspirated thrombotic material
3. LSFM and micro-CT for the assessment of the resected aortic valves. Finally, the scanned specimens will be histopathologically assessed at the First Department of Pathology in Athens, Greece by experienced pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Patients with sudden cardiac death for coronary artery imaging.
* Patients with STEMI undergoing PCI and thrombus aspiration for thrombus imaging.
* Patients with CAVD undergoing cardiac replacement of calcific aortic valve for valve imaging.

Exclusion Criteria:

* Patients dying after the execution of their cardiac surgery.
* Patients with altered mental status; unable or unwilling to provide informed consent for specimen imaging and clinical follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 cadaveric coronary artery segments with advanced atherosclerosis will be received from 10 patients with SCD who are likely to have advanced atherosclerosis. Additionally, 30 thrombotic specimens will be aspirated from patients presenting with STEMI. Finally, 30 aortic valves will be surgically removed from patients with CAVD undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Non-destructive nature of the deployed imaging modalities (Number of specimens with scanning-induced alterations) | 2 years
  The primary study outcome is to demonstrate the feasibility of ex vivo imaging of the collected cardiac specimens. Specifically, OCT, IVUS, LSFM and micro-CT will be used to scan cadaveric coronary arteries and the researchers will investigate that they can non-destructively image those specimens. Micro-CT will also be used for thrombotic material assessment and aortic valve imaging. Post-scanning histopathological assessment will be performed to confirm the non-destructiveness of the deployed imaging modalities and identify any radiation-induced or ischemic alterations within the scanned specimens.
Successful 3D visualization of the scanned specimens (generation of 3D datasets) | 2 years
  Co-primary study aim is to successfully scan all the collected specimens and produce 3D projections of the scanned specimens (i.e., 3D datasets).

SECONDARY OUTCOMES:
Micro-CT based quantification of the density (IU) within the scanned specimens | 2 years
  Quantitative density-related information will be received from micro-CT scanning of the 1) atherosclerotic plaques within the cadaveric coronary artery segments; 2) aspirated thrombotic samples; and 3) resected aortic valves (the measured density will represent the calcification).
Micro-CT based volumetric quantification (mm3) of the scanned specimens | 2 years
  Quantitative volumetric information can be received from micro-CT scanning of the 1) atherosclerotic plaque volume within the cadaveric coronary artery segments; 2) aspirated thrombotic volume; and 3) resected aortic valve volume.
Correlation of the derived images with histopathological data and visualization of regions of interest | 2 years
  The derived scans will be co-registered with the digital images (sections) generated by the histopathological assessment. IVUS, OCT, micro-CT and LSFM images will be matched to histopathological images (with immunohistochemistry and immunofluorescence analyses also performed). This might enable the identification of regions of interest (ROI) within the artery segments (intima, lipid-rich plaques and thrombi), the thrombotic specimens (red/white thrombus, WBC, platelets, hemosiderin) and the aortic valves (valvular cusps, amyloid, collagen and elastic fibers, valve annulus, leaflet and rest anatomic components).
Between-modality comparison of the image resolution achieved | 2 years
  Minimum voxel size and maximum resolution will be recorded and compared among the different imaging modalities, where applicable.
Between-modality comparison of the time required for image acquisition | 2 years
  Scanning and post-scanning reconstruction time will be recorded and compared among the different imaging modalities, where applicable.
IVUS-based quantification of areas of interest (mm2) within the scanned cadaveric arteries | 2 years
  Specific measurements of coronary areas of interest (Minimum lumen area, Lumen area stenosis, and Plaque area) will be derived from IVUS scanning of the cadaveric coronary artery segments.
IVUS-based quantification of diameters of interest (mm) within the scanned cadaveric arteries | 2 years
  Specific measurements of diameters of interest (Minimum lumen diameter, largest reference lumen diameter and distance from the distal to proximal reference site) will be derived from IVUS scanning of the cadaveric coronary artery segments.
IVUS-based determination of plaque characteristics within the scanned cadaveric arteries | 2 years
  Specific plaque characteristics will be determined (Plaque burden and Plaque type: Thick-cap fibroatheroma, Fibrotic plaque or Fibrocalcific plaque) through IVUS scanning of the cadaveric coronary artery segments.
IVUS-based determination of thrombotic characteristics within the scanned cadaveric arteries | 2 years
  If any thrombi are identified within the cadaveric coronary artery segments through IVUS scanning, thrombus characteristics will be determined according to the existing classification: 1) Acute thrombus (having an acoustic in-homogenous bright 'spontaneous contrast' appearance with sharp delineation and no clear signal attenuation), 2) Subacute thrombus (having a more homogeneous acoustic appearance and thus appearing darker), and 3) Organized thrombus (being the most acoustic homogeneous type of thrombus).
IVUS-based quantification of the thrombus score within the scanned cadaveric arteries | 2 years
  The thrombus score (derived from the SPECTRUM trial) will be calculated with IVUS scanning of the cadaveric coronary artery segments: 1-point adjudication for a total thrombus length >14.5 mm, 1-point for occlusive thrombus length >1.5 mm and 1-point for maximum thrombus angle 260°; this will be summarized as low (0-1 points) and high (2-3 points) thrombus burden.
OCT-based quantification of the assessed pathologies within the scanned cadaveric arteries | 2 years
  Specific measurements will be derived from OCT (attenuation coefficients for intimal tissue, lipid-rich tissue and thrombus) after scanning the cadaveric coronary artery segments.
LSFM-based quantification of the full-width half-maximum (FWHM) within the scanned cadaveric arteries | 2 years
  The FWHM of the light-sheet thickness will be calculated in the Z- and -Y directions, after scanning the cadaveric coronary artery segments.
LSFM-based quantification of the confocal parameter within the scanned cadaveric arteries | 2 years
  The confocal parameter will be calculated from LSFM scanning of the cadaveric coronary artery segments.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios I Tagarakis, MD, PhD, Principal Investigator — Cardiothoracic Surgery Department, Aristotle University of Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papazoglou AS, Karagiannidis E, Liatsos A, Bompoti A, Moysidis DV, Arvanitidis C, Tsolaki F, Tsagkaropoulos S, Theocharis S, Tagarakis G, Michaelson JS, Herrmann MD. Volumetric Tissue Imaging of Surgical Tissue Specimens Using Micro-Computed Tomography: An Emerging Digital Pathology Modality for Nondestructive, Slide-Free Microscopy-Clinical Applications of Digital Pathology in 3 Dimensions. Am J Clin Pathol. 2023 Mar 13;159(3):242-254. doi: 10.1093/ajcp/aqac143. PMID 36478204
- [Background] Papazoglou AS, Karagiannidis E, Moysidis DV, Sofidis G, Bompoti A, Stalikas N, Panteris E, Arvanitidis C, Herrmann MD, Michaelson JS, Sianos G. Current clinical applications and potential perspective of micro-computed tomography in cardiovascular imaging: A systematic scoping review. Hellenic J Cardiol. 2021 Nov-Dec;62(6):399-407. doi: 10.1016/j.hjc.2021.04.006. Epub 2021 May 12. PMID 33991670
- [Background] Karagiannidis E, Papazoglou AS, Sofidis G, Chatzinikolaou E, Keklikoglou K, Panteris E, Kartas A, Stalikas N, Zegkos T, Girtovitis F, Moysidis DV, Stefanopoulos L, Koupidis K, Hadjimiltiades S, Giannakoulas G, Arvanitidis C, Michaelson JS, Karvounis H, Sianos G. Micro-CT-Based Quantification of Extracted Thrombus Burden Characteristics and Association With Angiographic Outcomes in Patients With ST-Elevation Myocardial Infarction: The QUEST-STEMI Study. Front Cardiovasc Med. 2021 Apr 21;8:646064. doi: 10.3389/fcvm.2021.646064. eCollection 2021. PMID 33969012
- [Background] Karagiannidis E, Papazoglou AS, Stalikas N, Deda O, Panteris E, Begou O, Sofidis G, Moysidis DV, Kartas A, Chatzinikolaou E, Keklikoglou K, Bompoti A, Gika H, Theodoridis G, Sianos G. Serum Ceramides as Prognostic Biomarkers of Large Thrombus Burden in Patients with STEMI: A Micro-Computed Tomography Study. J Pers Med. 2021 Jan 31;11(2):89. doi: 10.3390/jpm11020089. PMID 33572568